CLINICAL TRIAL: NCT04690062
Title: Brolucizumab-dbll (BEOVU®) Intravitreal Injection in the Treatment of Dystrophy-related Macular Neovascular Degeneration
Brief Title: BEOVU in the Treatment of Dystrophy-related Macular Neovascular Degeneration
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, Lecturer of ophthalmology, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hamaky7
Record Dates: First submitted 2020-12-21; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Dystrophy, Retinal
Keywords: macular degeneration; BEOVU; RETINAL DYSTROPHY
MeSH Terms: conditions — Retinal Dystrophies; Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BEOVU (Experimental): Intravitreal injection of BEOVU 3 loading injections ( monthly) then every 3 months
  Interventions: Drug: Brolucizumab-Dbll

INTERVENTIONS:
Drug: Brolucizumab-Dbll — intravitreal injection of Brolucizumab (BEOVU)
  Other Names: BEOVU

SUMMARY:
Dystrophy-Related macular neovascularization degeneration occur is a vision threatening condition.The investigators evaluate the efficacy of BEOVU intravitreal treatment.

DETAILED DESCRIPTION:
Baseline ,and postoperative 1 ,6 and 12 months full ophthalmic examination was done.

Procedure included intravitreal injection of Brolucizumab (BEOVU®, Genen-tech, South Francisco, CA)

ELIGIBILITY:
Inclusion Criteria:

* Dystrophy-Related macular neovascularization degeneration

Exclusion Criteria:

* age related macular degeneration , other causes of macular neovascularization degeneration

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-25 (Actual); Primary Completion 2022-12-25 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity (BCVA) | 12 months
  Change in BCVA in LOG MARS(logarithm minimum angle of resolution)

SECONDARY OUTCOMES:
optical coherence tomography (OCT) foveal thickness | 12 months
  change in foveal thickness measured in micrometer

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Elhamaky, MD, Principal Investigator — Benha university faculty of medicine , INMC
Locations (1):
- INMC, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
by direct contact through email
Supporting Information: Study Protocol, SAP
Time Frame: unlimited
Access Criteria: direct request by email